CLINICAL TRIAL: NCT04439357
Title: MATCH Treatment Subprotocol S2: Phase II Study of Trametinib in Patients With Tumors With GNAQ or GNA11 Mutations
Brief Title: Testing Trametinib as a Potential Targeted Treatment in Cancers With GNAQ or GNA11 Genetic Changes (MATCH-Subprotocol S2)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03436; NCI-2020-03436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-S2 (Other: ECOG-ACRIN Cancer Research Group); EAY131-S2 (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (trametinib) (Experimental): Patients receive trametinib dimethyl sulfoxide PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Trametinib Dimethyl Sulfoxide

INTERVENTIONS:
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras

SUMMARY:
This phase II MATCH treatment trial identifies the effects of trametinib in patients whose cancer has genetic changes called GNAQ or GNA11 mutations. Trametinib may block proteins called MEK1 and MEK2, which may be needed for cancer cell growth when GNAQ or GNA11 mutations are present. Researchers hope to learn if trametinib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive trametinib dimethyl sulfoxide (trametinib) orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have GNAQ or GNA11 mutations, or another aberration, as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have NONE of the following cardiac criteria:

  * Clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
* Patients must have an echocardiogram (ECHO) or a nuclear study (multigated acquisition scan [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have a left ventricular ejection fraction (LVEF) < the institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients who previously received monoclonal antibody therapy (e.g., ipilimumab, nivolumab, pembrolizumab and others) must have stopped the prior therapy for 8 or more weeks before starting on trametinib
* Patients with glioblastoma must have histologically or radiographically confirmed recurrent or progressive World Health Organization (WHO) grade 4 glioma (glioblastoma).

  * NOTE: All baseline and post-baseline disease assessments must be performed using contrast-enhanced cranial magnetic resonance imaging (MRI) or contrast-enhanced computed tomography (CT) for subjects who cannot have MRI performed

Exclusion Criteria:

* Patients with a history of interstitial lung disease or pneumonitis are excluded
* Patients must not have known hypersensitivity to trametinib or compounds of similar chemical or biologic composition or to dimethyl sulfoxide (DMSO)
* Patients must not have a history or current evidence/risk of retinal vein occlusion (RVO). An eye exam is required at baseline
* Patients who previously received prior treatment with other MEK inhibitors (including, but not limited to, trametinib, binimetinib, cobimetinib, selumetinib, RO4987655 [CH4987655], GDC-0623 and pimasertib) will be excluded
* Patients with uveal melanoma are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Luke, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven patients were assigned to Subprotocol S2, 6 from screening cohort and 1 from outside laboratory. Of the 7 patients, 4 patients were enrolled in arm S2 between July 2016 and January 2019.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol S2, patients had to have a qualifying GNAQ or GNA11 actionable mutation.
Groups:
- Treatment (Trametinib): Patients receive trametinib dimethyl sulfoxide 2mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Trametinib Dimethyl Sulfoxide: Given PO
Period: Overall Study
Arm/Group | Treatment (Trametinib)
Started | 4
Eligible and Started Protocol Therapy (This is the primary analysis population.) | 4
Completed | 0
Not Completed | 4
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 62 [54 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for the detailed definitions of response criteria. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 4
percentage of participants | 25 [1.3 to 75.1]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 4
percentage of participants | 50 [22 to 100]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 4
months | 6.5 [1.8 to NA] — Median PFS 90% CI upper bound could not be determined due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis and all patients received protocol treatment were included in the toxicity analysis
Arm/Group | Treatment (Trametinib)
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib) (N=4)
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib) (N=4)
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Allergic reaction (Immune system disorders) | 1
Skin infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Hypertension (Vascular disorders) | 2
Lymphedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT04439357/Prot_001.pdf